CLINICAL TRIAL: NCT07062536
Title: A Randomized Phase II Clinical Trial to Evaluate the Efficacy Alternating mFOLFOX/mFOLFIRI Chemotherapy Regimen as a Second-line Treatment for Advanced Biliary Tract Cancer
Brief Title: mFOLFOX/mFOLFIRI vs. mFOLFOX in Advanced or Recurrent Biliary Tract Cancer Second-line
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jin Won Kim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Art-BTC
Record Dates: First submitted 2025-02-20; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Biliary Cancer Metastatic
Keywords: second line; alternating mFOLFOX/mFOLFIRI chemotherapy regimen
MeSH Terms: interventions — Oxaliplatin; Fluorouracil; Leucovorin; Irinotecan

STUDY DESIGN:
Intervention Model Description: Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mFOLFOX (Experimental): 1) mFOLFOX (Administered as a single regimen every 2weeks) D1 Oxaliplatin 85mg/m2 over 2hr Leucovorin 400mg/m2 over 2hr Fluorouracil 400mg/m2 FU 2400mg/m2 over 46hr
  Interventions: Drug: Oxaliplatin, 5FU, leucovorin
- mFOLFOX/mFOLFIRI (Experimental): (Administered alternately every 2 weeks.)
  1. mFOLFOX D1 Oxaliplatin 85mg/m2 over 2hr Leucovorin 400mg/m2 over 2hr Fluorouracil 400mg/m2 FU 2400mg/m2 over 46hr
  2. mFOLFIRI D1 Irinotecan 150mg/m2 over 2hr Leucovorin 100mg/m2 over 2hr 5FU 2400mg/m2 over 46hr
  Interventions: Drug: Oxaliplatin, 5FU, leucovorin/Irinotecan , 5FU, leucovorin,

INTERVENTIONS:
Drug: Oxaliplatin, 5FU, leucovorin — Administered as a single regimen every 2weeks
  Other Names: mFOLFOX
  Arms: mFOLFOX
Drug: Oxaliplatin, 5FU, leucovorin/Irinotecan , 5FU, leucovorin, — Administered alternately every 2weeks
  Other Names: mFOLFOX/mFOLFIRI
  Arms: mFOLFOX/mFOLFIRI

SUMMARY:
In second line with advanced or recurrent biliary tract cancer refractory to first line gemcitabine plus cisplatin,efficacy of mFOLFOX/FOLFIRI vs mFOLFOX will be evaluated at randomized phase 2 trial.

DETAILED DESCRIPTION:
1. brief enrollment criteria

   * histological confirmed
   * refractory to first line gemcitabine plus cisplatin
   * fit for chemotherapy
2. treatment arm A. mFOLFOX (Administered as a single regimen every 2weeks) 1) mFOLFOX D1 Oxaliplatin 85mg/m2 over 2hr Leucovorin 400mg/m2 over 2hr Fluorouracil 400mg/m2 FU 2400mg/m2 over 46hr

   treatment arm B. mFOLFOX/mFOLFIRI (Administered alternately every 2 weeks.) 1) mFOLFOX D1 Oxaliplatin 85mg/m2 over 2hr Leucovorin 400mg/m2 over 2hr Fluorouracil 400mg/m2 FU 2400mg/m2 over 46hr 2) mFOLFIRI D1 Irinotecan 150mg/m2 over 2hr Leucovorin 100mg/m2 over 2hr 5FU 2400mg/m2 over 46hr
3. randomization - stratified by site and performance status

   * Previous cancer treatment (including IO agents vs. excluding IO agents)

ELIGIBILITY:
Inclusion criteria (All eligibility criteria must be fulfilled)

1. Age ≥ 19 years.
2. Diagnosed with biliary tract cancer, including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, gallbladder cancer, or ampulla of Vater cancer.
3. Either unresectable advanced disease or recurrence after curative surgery.
4. ECOG (Eastern Cooperative Oncology Group) performance status of 0-2
5. First-Line Treatment Failure: Disease progression after at least one cycle of gemcitabine/cisplatin-based therapy or discontinuation of therapy due to adverse effects.
6. Presence of evaluable or measurable lesions according to RECIST v1.1 criteria.
7. Laboratory Criteria: optima bone marrow, liver, and kidney function within one week prior to enrollment: A. Hemoglobin > 9.0 g/dL B. Absolute neutrophil count (ANC) > 1,000/uL C. Platelet count > 75,000/uL D. Serum creatinine < 1.5× upper limit of normal (ULN) E. AST/ALT < 3× ULN F. Total bilirubin < 1.5× ULN (biliary drainage is allowed).
8. Patients who understand the study protocol, can provide written informed consent, and are aware of their right to withdraw at any time without penalty.
9. Effective Contraception (for patients of childbearing potential receiving oxaliplatin):

A. Male patients:

Must use effective contraception during the study and for 12 months after treatment completion.

B. Female patients:

Must use effective contraception during the study and for 15 months after treatment completion.

*Exclusion Criteria (Patients meeting any of the following criteria will be excluded from the study.)

1. Patients with prior exposure to oxaliplatin or irinotecan in previous cancer treatments.
2. Patients with metastatic or unresectable biliary tract cancer who have received second- line or higher chemotherapy.
3. Pregnant or breastfeeding women.
4. Patients with a history of other malignancies within the past 3 years, except for papillary or follicular thyroid cancer.
5. Patients with uncontrolled infections or other systemic diseases.
6. Patients with a history of myocardial infarction, unstable angina, or heart failure (NYHA
7. Class III-IV) within the last 6 months.
8. Patients with Grade 3 or higher peripheral neuropathy caused by prior chemotherapy.
9. Patients with known allergic reactions to the investigational drugs.
10. Known patients with Gilbert's syndrome, DPD (dihydro-pyrimidine dehydrogenase) deficiency, or Homozygous UGT1A1*28 alleles.
11. Patients currently taking potent CYP3A4 inhibitors (e.g., ketoconazole, itraconazole, ritonavir, clarithromycin), or potent CYP3A4 inducers (e.g., rifampin, carbamazepine, St.

    John's Wort).
12. Patients who are eligible for targeted therapy, including FGFR inhibitors or IDH1 inhibitors. (eligible for patient who unable to use these targeted agents due to drug cost.)
13. Patients with active CNS metastases and/or carcinomatous meningitis.
14. Patients who meet contraindications for the investigational drugs as per domestic regulatory guidelines, including patients with infections, Interstitial pneumonitis or pulmonary fibrosis, Severe diarrhea, Chronic inflammatory bowel disease, Intestinal paralysis or obstruction, Functional impairment due to peripheral sensory neuropathy, Severe renal dysfunction.
15. Patients deemed ineligible by the investigator for any other reason.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
6months overall survival rate | 6months
  at 6months from intervention treatment, overall survival rate

SECONDARY OUTCOMES:
response rate | 6months
  complete response,partial response
disease control rate | 6month
  complete response, partial response, stable disease
progression free survival | 6month
  from treatment start to progression or any cause of death
Number of participants with Treatment-Related Adverse Events as Assessed by NCI CTC version 4.0 | 6month
  percentage of all patients

CONTACTS AND LOCATIONS:
Overall Officials: Sun A Han, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Jin Won Kim, Seongnam-si, Out of US, South Korea

IPD SHARING:
Plan to Share IPD: No
The study does not explicitly state that patients with dementia or impaired renal function are to be enrolled according to the inclusion/exclusion criteria. However, based on exclusion criterion #14, "Others deemed inappropriate by the investigator," such patients cannot be enrolled.

DOCUMENTS (1):
  • Study Protocol (2025-01-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT07062536/Prot_000.pdf